CLINICAL TRIAL: NCT06646627
Title: Phase I Clinical Trial of Autologous B7-H3 Chimeric Receptor (CAR) T Cells in Adults With Recurrent, Platinum Resistant Ovarian Tumors
Brief Title: Clinical Trial of Autologous B7-H3 CAR T Cells in Reoccurent Platinum-resistant Ovarian Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-75080; NCI-2025-00266 (Registry Identifier: National Cancer Institute Clinical Trials Reporting Program)
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Ovarian Cancer
Keywords: B7-H3CART
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intraperitoneal (IP) Administration (Experimental): At the time of enrollment, based on imaging studies, clinical history and physical exams, the principal investigator will make a preliminary decision regarding Arm Assignment.
  Participants with ovarian cancer confined to the peritoneum will undergo laparoscopic placement of an intraperitoneal catheter (PowerPort™ device and catheter) for cell infusion. When feasible, a Tenckhoff catheter for research sample collection of ascites, will also be placed. If laparoscopic placement is not possible, the PowerPort catheter may be inserted in interventional radiology. If adhesions within the peritoneum would preclude effective distribution of CAR cells throughout the peritoneum, the participant may be placed in Arm B.
  Interventions: Drug: B7-H3CART
- Intravenous (IV) Administration (Experimental): At the time of enrollment, based on imaging studies, clinical history and physical exams, the principal investigator will make a preliminary decision regarding Arm Assignment.
  Arm B will consist of participants with disease outside the peritoneum and with participants who either cannot undergo IP catheter insertion or who, in the judgement of the principal investigator do not have an intraperitoneal environment that would allow for adequate product distribution. Participants in Arm B will have a Tenckhoff catheter inserted in Interventional Radiology at least 7 days before the start of conditioning lymphodepletion.
  Interventions: Drug: B7-H3CART

INTERVENTIONS:
Drug: B7-H3CART — Dose Levels:
  Dose Level -1 Dose Level 1 Dose Level 2 Dose Level 3
  Arm A IP(± 20%) (flat dose) Dose Level -1: 1 x 107 B7-H3CART Dose Level 1: 5 x 107 B7-H3CART Dose Level 2: 15 x 107 B7-H3CART Dose Level 3: 5 x 108 B7-H3CART
  Arm B: IV (± 20%) (weight based) Dose Level -1: 3 x 105 transduced cells/kg Dose Level 1: 1 x 106 transduced cells/kg Dose Level 2: 3 x 106 transduced cells/kg Dose Level 3: 10 x 106 transduced cells/kg

SUMMARY:
This is a single site, open label, Phase 1 study using a 3 + 3 dose escalation design in two cohorts of adults with recurrent, platinum-resistant ovarian tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Disease: Histologically or cytologically confirmed diagnosis of ovarian cancer including serous, endometrioid, clear cell, mucinous, mixed epithelial, or undifferentiated. The study does not include pure sarcoma, stromal, or germ-cell tumors. Tumors that are substantially high-grade carcinoma and have focal elements of lower grade tumors or sarcomatous elements (e.g., carcinosarcoma) are eligible.
2. Have measurable disease. Measurable disease is defined as at least 1 lesion that can be accurately measured in at least 1 dimension (longest diameter to be recorded). Each lesion must be ≥10 mm when measured by CT, MRI, or caliper measurement at clinical examination or ≥20 mm when measured by chest x-ray. Lymph nodes must be ≥15 mm in short axis when measured by CT or MRI.
3. B7-H3 positive expression on malignant cells is NOT required but archival tissue must be available, or the subject must be willing to undergo tissue biopsy for expression analysis.
4. Age: ≥ 18 years of age
5. Prior Therapies: Subjects must have had at least 1 prior platinum-based chemotherapeutic regimen for the management of ovarian carcinoma.

   Patients should be considered platinum- refractory (progression while on a prior platinum chemotherapy) or resistant (persistence or recurrence within 6 months after a prior platinum-based chemotherapy) after all available curative standard therapies. There is no limit to the number of prior therapies.

   At least 3 weeks post chemotherapy or 5 half-lives, whichever is shorter, must have elapsed since any prior systemic therapy, except for systemic inhibitory/stimulatory immune checkpoint therapy that requires 3 months.

   Must have recovered from prior therapy toxicities to grade 1 or baseline, except for peripheral neuropathies, alopecia, etc.
6. Performance Status: ECOG status of 2 or better (or Karnofsky Performance Status score of ≥60%) (See Section 11.1)
7. Life expectancy at least 3 months, in the investigator's clinical judgement.
8. Adequate bone marrow and major organ function.

   * Hgb ≥ 10 g/dL
   * ANC ≥ 1500/uL
   * Platelet count ≥ 100,000/uL
   * Absolute lymphocyte count ≥150/uL
   * Creatinine ≤ 1.5 mg/dL or creatinine clearance ≥ 50 mL/min
   * Serum ALT and AST ≤ 5x ULN (Grade 2)
   * Total bilirubin ≤ 1.5x ULN (subjects with Gilbert's syndrome allowed if direct bilirubin within normal limits)
   * PT or PTT ≤ 1.25 X ULN (not receiving therapeutic anticoagulation)
   * Cardiac ejection fraction ≥ 45%
   * No evidence of physiologically significant pericardial effusion
   * No clinically significant ECG findings
   * Baseline oxygen saturation > 92% on room air
9. Pregnancy: Females of childbearing potential (defined as women ≤50 years of age, or >50 years of age with a history of amenorrhea for ≤12 months prior to study entry) must have a negative blood or urine pregnancy test.

Subjects of child bearing potential must be willing to use an effective method of contraception (hormonal or two barrier methods) from the time of enrollment on this study and for at least four (4) months after receiving last dose of B7-H3CART cells or until CAR T cells are undetectable in peripheral blood.

10. Consent: Must be able to understand and be willing to personally sign the written IRB approved informed consent document.

Exclusion Criteria:

* 1. Active infection or uncontrollable infection requiring systemic treatment within 1 week before screening. Simple UTI and uncomplicated bacterial pharyngitis are permitted if responding to active treatment.

  2. Requirement for systemic corticosteroid therapy at doses higher than physiologic maintenance dosing (must be < 5 mg/day of prednisone (or equivalent doses of other corticosteroids). Topical, inhaled or ocular steroids are allowed.

  3. Presence of abdominal fistula, gastrointestinal perforation, or intraabdominal abscess.

  4. Malignant tumors other than the target tumor within 2 years prior to screening, except for the following: malignant tumors that have received radical treatment and no known active disease within ≥ 2 years prior to enrollment; or adequately treated non-melanoma skin cancers with no evidence of disease.

  5. Have any of the following heart conditions:

  • New York Heart Association (NYHA) stage III or IV congestive heart failure;
  * Myocardial infarction or coronary artery bypass grafting (CABG) within 6 months before enrollment;
  * Clinically significant ventricular arrhythmia, or a history of unexplained syncope (except those caused by vasovagal or dehydration);
  * History of severe nonischemic cardiomyopathy. 6. Known to have active or uncontrolled autoimmune diseases, such as Crohns disease, rheumatoid arthritis, systemic lupus erythematosus, systemic vasculitis, etc.

    7. Ongoing HIV, HBV, or HCV infection. History of HBV or HCV is permitted if viral load is undetectable by qPCR and/or nucleic acid testing.

    8. Known or suspected untreated brain metastases. Patients with radiographically stable, asymptomatic previously irradiated lesions are eligible provided patient is >4 weeks beyond completion of cranial irradiation and >3 weeks off of corticosteroid therapy at the time of study intervention.

    9. Known sensitivities to any of the agents used in this study or their reagents including steroids, tocilizumab, DSMO, cyclophosphamide, fludarabine, etc.

    10. Prior history of clinically significant seizure disorder (e.g., not including childhood febrile seizures).

    11. Any other issue which, in the opinion of the treating physician or principal investigator, would make the patient ineligible for the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility of B7-H3CART Manufacturing | 2 years
  Feasibility is defined by the frequency of successful manufacturing runs of B7-H3CART that meet the established Investigational New Drug (IND) release criteria and the targeted dose level.
Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) | 28 days after B7-H3CART infusion
  MTD and/or RP2D defined in each arm (IP and IV) based on the number of events meeting definition of dose limiting toxicity (DLT) measured 28 days after infusion, tested in at least 6 evaluable participants in each arm.

SECONDARY OUTCOMES:
Number of Subjects Meeting RECIST Radiographic Response at Day 28 to Determine Response Rate (RR) and Duration of Response (DOR) | 12 months
  Number of subjects who meet RECIST radiographic response at Day +28 to determine Response rate (RR) and duration of response (DOR) at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Dorigo, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States